CLINICAL TRIAL: NCT02341508
Title: A Phase 1a, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Lpathomab Administered Intravenously to Healthy Volunteers
Brief Title: A Phase 1a, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate Lpathomab in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lpath, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT3114-NPP-001
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Saline Solution; Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lpathomab (Experimental): 0.5 mg/kg Lpathomab, 1.0 mg/kg Lpathomab, 3.0 mg/kg Lpathomab, 10 mg/kg Lpathomab, 20 mg/kg Lpathomab,
  Interventions: Biological: 0.5 mg/kg Lpathomab; Biological: 1.0 mg/kg Lpathomab; Biological: 3.0 mg/kg Lpathomab; Biological: 10 mg/kg Lpathomab; Biological: 20 mg/kg Lpathomab
- Placebo (Placebo Comparator): Saline solution for intravenous infusion
  Interventions: Other: Saline solution for intravenous infusion

INTERVENTIONS:
Biological: 0.5 mg/kg Lpathomab
  Arms: Lpathomab
Biological: 1.0 mg/kg Lpathomab
  Arms: Lpathomab
Biological: 3.0 mg/kg Lpathomab
  Arms: Lpathomab
Biological: 10 mg/kg Lpathomab
  Arms: Lpathomab
Biological: 20 mg/kg Lpathomab
  Arms: Lpathomab
Other: Saline solution for intravenous infusion
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of Lpathomab in healthy volunteers. Additional endpoints include characterization of the pharmacokinetic (PK), pharmacodynamic (PD), and immunogenicity profiles of a single IV dose of Lpathomab in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male or female subject ≥ 18 years old between 50 and 145 kg
* Laboratory values and ECG during Screening period within normal range or evaluated as not clinically significant (NCS)
* Female subjects must be not of child-bearing potential or using double-barrier method of contraception
* Male subjects must use double-barrier contraception during the study period
* Subject is able to read, understand, and sign the informed consent form (ICF) and HIPAA release

Key Exclusion Criteria:

* Subjects with diabetes mellitus (glycated hemoglobin [HbA1c]≥6.5%) or pre-diabetes mellitus (HbA1c between 5.7 and 6.4%).
* Male subjects with corrected Q-T interval (QTc)> 450 msec or a QRS interval>120 msec and female subjects with QTc> 470 or a QRS interval>120 msec.
* Subject's blood pressure (BP) during screening period exceeds 140/90 mm Hg
* Subject is positive for HIV, hep B and/or hep C at screening
* Subject has significant psychiatric co-morbidity including but not limited to major depression-severe, bipolar disorder or schizophrenia spectrum disorder, history of suicide attempt, or active suicidal ideation in 6 months prior to screen.
* Subject has any significant or advanced systemic illness, unstable or severe medical condition(s) or end stage disease that could put them at risk during the study, interfere with outcome measures, or affect compliance with the protocol procedures and requirements.
* Subject has history of cancer stability/remission for less than 5 years, with the exception of non-metastatic basal and/or squamous cell carcinomas of the skin and cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with local or systemic Adverse Events | 85 days

CONTACTS AND LOCATIONS:
Overall Officials: Dario A Paggiarino, MD, Study Director — Lpath, Inc.
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States